CLINICAL TRIAL: NCT00696969
Title: Randomized, Open-label, Parallel-group, Safety & Efficacy Study to Evaluate Different Combination Treatment Regimens, of Either AmBisome and Paromomycin, AmBisome and Miltefosine, or Paromomycin and Miltefosine Compared With Amphotericin B Deoxycholate (the Standard) Therapy for the Treatment of Acute, Symptomatic Visceral Leishmaniasis (VL).
Brief Title: Safety and Efficacy Study to Evaluate Different Combination Treatment Regimens for Visceral Leishmaniasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Responsible Party: Clinical Project Coordinator, DNDi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VL Combo 07
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2010-02-11 (Estimated); Status verified 2010-02

CONDITIONS: Visceral Leishmaniasis
MeSH Terms: conditions — Leishmaniasis, Visceral | interventions — amphotericin B, deoxycholate drug combination; liposomal amphotericin B; miltefosine; Paromomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator)
  Interventions: Drug: Amphotericin B Deoxycholate
- 2 (Experimental)
  Interventions: Drug: Ambisome + Miltefosine
- 3 (Experimental)
  Interventions: Drug: Ambisome and Paromomycin
- 4 (Experimental)
  Interventions: Drug: Miltefosine and Paromomycin

INTERVENTIONS:
Drug: Amphotericin B Deoxycholate — 1 mg/kg e.o.d for 30 days
  Arms: 1
Drug: Ambisome + Miltefosine — Ambisome (i.v. single dose 5 mg/kg)+ Miltefosine 7 days
  Arms: 2
Drug: Ambisome and Paromomycin — Ambisome 5 mg/kg single dose + Paromomycin Sulphate 15mg/kg/day for 10 days
  Arms: 3
Drug: Miltefosine and Paromomycin — Miltefosine (standard dose) and Paromomycin Sulphate 15mg/kg/day for 10 days
  Arms: 4

SUMMARY:
The overall objective of this trial is to identify a safe and effective combination, (coadministration) short course treatment for the treatment of visceral leishmaniasis which could be easily deployed in a control programme and will reduce the risk of parasite resistance occurring.

Safety and tolerability should be such that the combination can be easily deployed.

DETAILED DESCRIPTION:
New, effective, less toxic and simplified treatments are urgently needed to replace or complement the few currently available drugs to treat visceral Leishmaniasis. An interim strategy and one which will slow the emergence of resistant parasite strains is to use coadministration of currently available drugs.

In India, first line treatment is now amphotericin B which is administered as an intravenous infusion, on alternate days over a 4 week period. A liposomal formulation of amphotericin B, AmBisome, is also available, and is substantially less nephrotoxic than amphotericin B, but is expensive.

It is acknowledged that AmBisome is the most effective therapy for visceral leishmaniasis, but it's high cost has hampered implementation. Use as part of a combination treatment, potentially as a single, lower dose, could reduce treatment costs considerably and thereby increase access for patients.

Two new treatments have recently been licensed in India for the treatment of patients with VL,

* Paromomycin administered as an intramuscular injection, once daily for 21 days
* Miltefosine administered as an oral tablet, once daily for 28 days. These drugs are now being used as monotherapy with high risk of emergence of resistant parasites. With price reduction for AmBisome, preferential pricing for Miltefosine and the concern for emergence of resistant parasites due to monotherapy, it is time to move rapidly toward obtaining definitive data for making recommendations on combination therapy as soon as possible, before these valuable drugs become useless. The present protocol will be a definitive Phase-III trial with the aim that at the end of this trial, strong evidence-based recommendations on combination therapy with available drugs can be made to Authorities in the Indian sub-continent. This protocol will evaluate various combinations of the three drugs; AmBisome, Paromomycin and Miltefosine at reduced total dosage and in shorter courses, against the present standard treatment with amphotericin B deoxycholate.

ELIGIBILITY:
Inclusion Criteria:

* Adults ( male or female) 18-60 years of age
* Acute, symptomatic, non-severe (minimum Hb.5 gm/dL) VL proven by parasitological examination of splenic or bone marrow aspirate.
* History of fever.
* Living within reachable distance of the trial site to enable attendance for follow-up visits
* Written informed consent to participate
* Proven HIV negative status
* Women of child-bearing potential who are using an assured method of contraception

Exclusion Criteria:

* Signs/symptoms indicative of severe VL ( Hb.< 5gm/dl, evidence of cardiac failure, etc)
* Patients who have received anti-leishmanial or anti-fungal treatment within the last 45 days
* Patients who have received any investigational (unlicensed) drugs within the last 6 months
* Severe malnutrition BMI<15 in adults, weight for height less than 60% in children.
* Chronic underlying disease such as severe cardiac, renal, or hepatic impairment.
* Renal function tests (serum creatinine) outside the normal range
* Liver function tests (transaminases) more than three times the upper limit of the normal range at study entry
* Jaundice (bilirubin >2.0mg/dL)
* Known hepatitis B or C positive
* Platelet count less than 40,000/mm3
* Prothrombin time 5 seconds or greater than normal range
* TotalWBC < 1,000/mm3
* Known alcohol or other drug abuse
* HIV positive status
* Pregnancy and/or lactation
* Females having unprotected sexual intercourse, or using a non-assured method of contraception (e.g. condom)
* Concomitant chronic drug treatment eg for diabetes, hypertension, TB, HIV etc
* Concomitant drug usage for acute infection, eg malaria, pneumonia etc within the last 7 days
* Any other condition which may invalidate the trial
* Known hypersensitivity to AmBisome, Paromomycin, amphotericin B and/or Miltefosine

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 634 (Actual)
Dates: Start 2008-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Definitive cure based on parasitological clearance at Day 15 after start of combination therapy (Day 31 for standard therapy), no evidence of parasites at day 45 and no clinical signs or symptoms of VL at 6 months post treatment. | 6 months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Farrokh Modabber, Study Director — Drugs for Neglected Diseases
Locations (2):
- India (2):
  - Kala-azar medical centre, Muzaffarpur, Bihar
  - Rajendra Memorial research Institute, Patna, Bihar

REFERENCES:
- [Derived] Sundar S, Sinha PK, Rai M, Verma DK, Nawin K, Alam S, Chakravarty J, Vaillant M, Verma N, Pandey K, Kumari P, Lal CS, Arora R, Sharma B, Ellis S, Strub-Wourgaft N, Balasegaram M, Olliaro P, Das P, Modabber F. Comparison of short-course multidrug treatment with standard therapy for visceral leishmaniasis in India: an open-label, non-inferiority, randomised controlled trial. Lancet. 2011 Feb 5;377(9764):477-86. doi: 10.1016/S0140-6736(10)62050-8. Epub 2011 Jan 20. PMID 21255828